CLINICAL TRIAL: NCT05803213
Title: Learning Efficacy and Motivation of Medical Students Between Different Teaching Materials and Methods in Clinical Training for Anesthesia and Perioperative Care
Brief Title: Learning Efficacy and Motivation of Medical Students in Clinical Training With Virtual Reality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 202201058RINA
Record Dates: First submitted 2023-03-15; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Motivation; Efficacy, Self

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The assessors do not know the group assignment. The investigators who handle data analysis and statistics do not know the group assignment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (Experimental): The medical students use the virtual reality headset to watch an interactive 360 video about the clinical situation on the learning platform
  Interventions: Other: Virtual Reality 360 interactive video
- Traditional (Active Comparator): The mini-lecture is provided by the instructor to medical students about the clinical situation
  Interventions: Other: Traditional mini-lecture

INTERVENTIONS:
Other: Virtual Reality 360 interactive video — Clinical scenarios revised and presented with 360 video, and interactive design on the learning platform that is available anytime and anywhere to the medical students
  Arms: Virtual Reality
Other: Traditional mini-lecture — Clinical scenario described according to the script as a mini-lecture to the medical students
  Arms: Traditional

SUMMARY:
We created a curriculum based on clinical events with 360° camera on an interactive learning platform. We hypothesize that medical students will learn better and be motivated with the immersive 360 video and virtual reality headset during the clinical training.

DETAILED DESCRIPTION:
We created a curriculum based on rapid sequence induction before anesthesia induction with 360° camera and put it on an interactive learning platform. We hypothesize that medical students will have better learning efficacy and motivation with the immersive 360 video and virtual reality headset. Moreover, the learning engagement will be translated into clinical skills acquisition and medical knowledge retention.

ELIGIBILITY:
Inclusion Criteria:

* Medical students undergoing clinical rotation

Exclusion Criteria:

* Unable to wear virtual reality headset

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Learning Efficacy | 6 months
  Learning Efficacy that is assessed by questionnaire
Learning Motivation | 6 months
  Learning Motivation that is assessed by questionnaire

SECONDARY OUTCOMES:
Clinical skills | 6 months
  Clinical skills associated with the clinical scenario that are assessed by simulation on a phantom and checklists

OTHER OUTCOMES:
Medical knowledge | 6 months
  Medical knowledge associated with the clinical scenario that is assessed by written tests

CONTACTS AND LOCATIONS:
Overall Officials: Man-Ling Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis."
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 9 months after article publication for up to 24 months
Access Criteria: Access to trial data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact the principle investigator